CLINICAL TRIAL: NCT02715921
Title: Impact of Telerehabilitation Training on Pediatric Cystic Fibrosis Patients: An Exploratory Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 277-13
Record Dates: First submitted 2016-01-12; First posted 2016-03-22 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cystic fibrosis patients (Experimental): Receive tele-exercise training and undergo pulmonary function testing and exercise testing
  Interventions: Other: Tele-exercise

INTERVENTIONS:
Other: Tele-exercise

SUMMARY:
Fitness in patients with Cystic fibrosis (CF) is an important biomarker associated with higher survivability and improved quality of life. CF patients are encouraged to maintain an active lifestyle, however, while physicians are able to prescribe airway clearance measures or specific medications, there is no prescription for exercise or avenue to promote exercise outside the clinic or hospital.

DETAILED DESCRIPTION:
The advent of ubiquitous computing has transformed the landscape of healthcare delivery. Thus far, exercise training in CF have either required patients travel to a gym or relied on home visits or telephone calls. Virtual visits provide a novel and innovative platform to deliver a live stream of exercise sessions with two-way video and audio capabilities, allowing individualized attention to exercise for CF patient from the comfort and privacy of their homes. Applications of tele-exercise, or tele-rehabilitation, have been shown to be as effective as in conventional physical therapy following orthopedic surgeries and, in stroke patients, to optimize patient outcome by prolonging duration of treatment and preventing the observed decline after the termination of therapy. For CF patients, the latter is especially important given the impact of hospitalizations for acute exacerbations on exercise tolerance. In this particular population, where cross-contamination risks limit use of group exercise activity, using two-way video telecommunication allows participation in exercise programs while adhering to the standards of CF management regarding infection control.

This study would be the first to evaluate implementing tele-exercise and remote monitoring program on pediatric CF patients. Pediatric CF patients will be enrolled in a six-week exercise program that is streamed live from an instructor into their computers at home via a HIPAA compliant telemedicine platform. Remote monitoring devices, such as accelerometers and wireless heart rate monitors, will evaluate baseline habitual activity and intensity of exercise, respectively. The goal of this study is to show that tele-exercise program is a feasible and convenient and cost-effective method to enhance CF care.

ELIGIBILITY:
Inclusion Criteria

* 8 - 21 years old
* Diagnosis of Cystic Fibrosis confirmed by genetic studies and/or sweat chloride testing
* Baseline pulmonary function testing (PFT) (within the last 3 months) with FEV1 (Forced expiratory volume in 1 second) > 40%
* Must be able to perform 3-minute step test.
* Must achieve an adequate 15 count breathlessness score. Must be able to perform ergometry testing utilizing extremities
* Must have a working computer/smartphone/tablet with internet connection at home

Exclusion criteria

* FEV1 < 40%
* Desaturations (less than 75%) or significant fatigue with 3-minute step test 15 count breathlessness score of greater than 2
* Pulmonary exacerbation (shortness of breath or difficulty breathing requiring hospitalization) within the last 4 weeks
* Oxygen requirement at rest or during sleeping.
* Recent pneumothorax (popped lung) within last 3 months
* Moderate pulmonary hypertension (increased pressure in the lung arteries) diagnosed via echocardiogram.
* History of low ejection fraction (percentage of blood being pumped out of the heart) via echocardiogram.
* History of cardiac ischemia (reduced blood supply to heart tissue).
* Uncontrolled systemic hypertension for patient age and height.
* Moderate to severe scoliosis (abnormal curvature of the spine)

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Habitual activity | 7 days
  An Actigraph accelerometer will be worn by the participant during waking hours for the first week and last week of the exercise program to assess habitual activity.

SECONDARY OUTCOMES:
Peak oxygen consumption | 30 minutes
  The patient will exercise on a cycle ergometer, using a ramp protocol in which the resistance is increased by 10-20 watts per minute, until exhaustion. During this test, breath by breath measurements of physiological parameters (oxygen saturation, carbon dioxide levels, respiratory rate, heart rate) will be measured. From these measurements, we will extrapolate VO2 (oxygen consumption) at its peak, which is when the participant reaches his or her highest level of exertion.
Cystic fibrosis quality of life survey | 50 minutes
  Approximately 50 questions related to quality of life in Cystic fibrosis.
System usability survey | 10 minutes
  A ten question survey related to system usability. Answers for these questions range from 0 (strongly disagree) to 4 (strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Jen Jen Chen, MD, Principal Investigator — MemorialCare
Locations (1):
- Pediatric Exercise and Genomics Research Center, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No